CLINICAL TRIAL: NCT04976283
Title: Which Oral Combination of Anti-diabetes Medication May Work Better in Subjects With Type 2 Diabetes and Nonalcoholic Fatty Liver Disease: a Randomized Control Trial
Brief Title: Effect of Oral Anti-diabetic Medication on Liver Fat in Subjects With Type II Diabetes and Non-alcoholic Fatty Liver
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Getz Pharma (Industry)
Responsible Party: Principal Investigator, Dr. Najmul Islam, Professor Endocrinology, Diabetes, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKUH-GTZ-DM-005-21
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2; NASH - Nonalcoholic Steatohepatitis; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pioglitazone (Active Comparator): The starting dose would be 15mg/day for pioglitazone and 500 to 1500mg per day for metformin (depending on blood glucose levels). Starting dose for DPP4 inhibitors would be 50 to 100mg daily.
  Interventions: Drug: Pioglitazone
- Empagliflozin (Active Comparator): The starting dose would be 500-1500mg/day of metformin, plus 5/10/12.5mg empagliflozin (depending on blood glucose levels). Starting dose for DPP4 inhibitors would be 50 to 100mg daily.
  Interventions: Drug: Empagliflozin
- Pioglitazone + Empagliflozin (Active Comparator): The starting dose would be 15mg/day for pioglitazone and 500 to1500mg per day for metformin and 5/10/12.5mg/25mg/day empagliflozin and 50 to 100mg daily for DPP4 inhibitors depending on blood sugar levels.
  Interventions: Drug: Pioglitazone + Empagliflozin

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone with (or without) metformin and/or DPP4 inhibitor (no SGLT2 inhibitor). The maximum dose for metformin would be 2.5 g/day, while for pioglitazone would be 45mg/day. The maximum dose for DPP4 inhibitor would be 100mg/day.
  Other Names: Zolid
  Arms: Pioglitazone
Drug: Empagliflozin — Empagliflozin with (or without) metformin and/or DPP4 inhibitor (no pioglitazone). The maximum dose for metformin would be 2.5g/day, while for empagliflozin would be 25mg/day depending on follow up blood sugar levels and tolerability. The maximum dose 100mg daily.
  Other Names: Diampa
  Arms: Empagliflozin
Drug: Pioglitazone + Empagliflozin — Pioglitazone with (or without) metformin and/or DPP4 inhibitor, plus empagliflozin. The maximum dose for metformin would be 2.5g/day; for pioglitazone would be 45mg/day and 25mg/day for empagliflozin, and 100mg daily for DPP4 inhibitors (depending on follow up blood sugar levels and tolerability).
  Other Names: Zolid + Diampa
  Arms: Pioglitazone + Empagliflozin

SUMMARY:
This randomized clinical trial aims to compare the effect of the pioglitazone and SGLT2 inhibitor combination on liver fat mass, as compared to either drug used alone, with or without background medical therapy of metformin and/or DDP4 inhibitors.

DETAILED DESCRIPTION:
To compare the effect of pioglitazone with or without Metformin and/or DPP4 inhibitor (no SGLT2 inhibitor) on improvement of NAFLD parameters, versus

The effect of SGLT inhibitor with or without metformin and/or DPP4 inhibitor (no pioglitazone) on NAFLD parameters and versus

Pioglitazone with or without metformin and/or DPP4 inhibitor, plus empagliflozin on improvement of NAFLD parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient who give informed consent voluntarily
* Type 2 diabetic patient having age from 18 years to 60 years
* HbA1C ≥ 7.0 %
* Diabetes diagnosis of ≤ 5 years (longer duration more likely to be associated with use of multiple drug regimens for glycemic control which may affect liver fat mass)
* Either treatment naïve or on metformin alone or metformin/DPP4i combination
* Absolute weight < 100kg; BMI < 45 (fibro scan machine cannot accommodate heavier individuals)
* Documented hepatosteatosis (If the fibroscan reveals S1 (mild fatty liver: 11-33% fatty liver) to S3 (severe fatty liver: > 67% fatty liver) liver fat

Exclusion Criteria:

* Hba1c ≥ 9% and/or blood sugar > 250mg/dl
* History of uncontrolled Endocrine disorder (for example uncontrolled hypothyroidism, or that requiring frequent dose adjustment, or Cushings syndrome)
* History of anti-obesity medication use within 3 months of consent for study enrollment or weight loss procedure(bariatric surgery) within same duration
* History of use of SGLT 2 inhibitors, glitazones, Glucagon-like peptide (GLP) 1 agonists 3 months prior to study enrollment as they influence liver fat
* History of use of insulin/sulphonylurea 3 months prior to study enrollment owing to weight gain and potential increase in liver fat conferred by these agents
* History of vitamin E use (400mg twice daily) within 3 months of study enrollment
* Drug induced liver disease or active substance abuse (cannabonnoid-derived substances like heroin, cocaine, amphetamines) based on history and/or laboratory tests
* Drugs known to be associated with hepatic steatosis like steroids, traditional homeopathic medication (likely to contain steroids), methotrexate, valproate, tamoxifen, amiodarone.
* Alcohol use (History of alcoholism or a greater than recommended alcohol intake (> 21 standard drinks on average per week in men and > 14 standard drinks on average per week in women)
* Severe hepatic impairment (ALT levels > 3 times upper limit normal)
* Hepatitis B/C hepatitis (based on positive Hepatitis B surface antigen, Anti Hepatitis C antibodies positive
* Autoimmune hepatitis (in case of females), based on positive Anti-nuclear Antibody (ANA) (homogenous, high titre)
* Positive Human Immunodeficiency Virus ( HIV) test as this could influence liver functions
* Pregnant or lactating women/ plans for pregnancy over proceeding 13 months
* Obstructive liver disease on the basis of laboratory and imaging studies
* Chronic renal failure, or Glomerular Filtration Rate (GFR) < 30 mls/minute (as estimated by the MDRD equation)
* Chronic heart failure, history of acute coronary artery disease or cerebrovascular accident within 3 months of consent for study enrollment, based on history and/or cardiac imaging
* History of recurrent Urinary Tract Infections (UTI's) or mycotic infections
* Presence of ketones on Urine Analysis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in radiologic liver parameters | 12 months
  Number of participants reported change in liver fat content from baseline, as quantified by fibroscan

SECONDARY OUTCOMES:
Change in liver enzymes | 12 months
  Number of participants reported change in liver enzymes levels including ALT, AST and GGT
Change in Fibrosis-4 (FIB-4) Score and NAFLD Fibrosis Score | 12 months
  Number of participants reported change in FIB-4 Score and NAFLD Fibrosis Score. Fibrosis-4 scores range from 0 to 4, where <1.45 indicates absence of cirrhosis; score between 1.45 - 3.25 are deemed inconclusive and score >3.25 indicates cirrhosis.
Change in body weight | 12 months
  Number of participants reported change in body weight from baseline (treat to target response of at least 5% of baseline at 6 months, 10% baseline over 12 months).
Change in waist circumference (WC) | 12 months
  Number of participants reported change in waist circumference (WC)
Change in liver fat mass with total body fat (TBF) | 12 months
  Comparison of baseline and end of treatment liver fat mass with total body fat (TBF) using a Body Composition Monitor
Change in HbA1C levels (< 7.0%) | 12 months
  Number of participants reported change in HbA1C levels from baseline to end of treatment
Change in Fasting Blood Sugar (FBS) | 12 months
  Number of participants reported change in Fasting Blood Sugar (FBS) from baseline to end of treatment
Change in Lipid profile | 12 months
  Number of participants reported change in Fasting triglycerides (TG), Low-Density Lipoprotein (LDL), High-Density Lipoprotein (HDL) from baseline to end of treatment

OTHER OUTCOMES:
Change in Urine Albumin to Creatinine Ratio (UACR) | 12 months
  Number of participants reported change in Urine Albumin to Creatinine Ratio (UACR) from baseline to end of treatment
Change in Systolic and Diastolic blood pressure | 12 months
  Number of participants reported change in Systolic and Diastolic blood pressure from baseline to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan